CLINICAL TRIAL: NCT03440294
Title: Étude de l'Effet de la Combinaison néoprène et de l'équipement Individuel de Flottaison Sur la Fonction Respiratoire de Repos et Les capacités à l'Effort Chez Les véliplanchistes : étude WINDSURF
Brief Title: Wetsuit and Life Jacket Induced Effects on Spirometry and VO2 in Windsurfers
Acronym: WINDSURF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC17.0233
Record Dates: First submitted 2018-01-31; First posted 2018-02-22 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Ventilation; Exercise
Keywords: windsurfer; wetsuit; spirometry; cardiopulmonary exercise testing; lung function; pulmonary function; oxygen uptake
MeSH Terms: conditions — Respiratory Aspiration; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with neoprene suit and life jacket (Other): Realization of the following examinations WITH neoprene suit and life jacket :
  * resting standard spirometry
  * maximum exercise testing. No drug and no placebo will be used in this arm.
  Interventions: Diagnostic Test: resting standard spirometry; Diagnostic Test: maximum exercise testing
- without neoprene suit and life jacket (Other): Realization of the following examinations WITHOUT neoprene suit and life jacket :
  * resting standard spirometry
  * maximum exercise testing. No drug and no placebo will be used in this arm.
  Interventions: Diagnostic Test: resting standard spirometry; Diagnostic Test: maximum exercise testing

INTERVENTIONS:
Diagnostic Test: resting standard spirometry — The subject (seated, bust straightened) should perform, after a slow and maximum inspiration, a forced and complete exhalation followed by a new inspiration to the total lung capacity.
Diagnostic Test: maximum exercise testing — Incremental exercise on cycle ergometer with 100W start for men (80W for women) for 4 minutes as part of the warm-up. Then, step increment of a 50W power for men (40W for women) lasting 2 minutes each.

SUMMARY:
The purpose of this study is to investigate the effect of wearing both neoprene suit and life jacket on respiratory capacities at rest and cardiopulmonary capacities during exercise in windsurfers.

DETAILED DESCRIPTION:
Windsurfers will perform resting spirometry and exercise test on cycle ergometer until exhaustion in two conditions: with or without equipment. The investigators will measure Forced Vital Capacity, FEV1 peak flow at rest and oxygen uptake, carbon dioxide consumption, ventilation at each step of the incremental exercise and at exhaustion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 35
* Do not contraindicate any of the investigations in the study
* Being affiliated to a social security system
* free, informed and written consent
* Have already performed a cardiopulmonary exercise test without any electrocardiographic abnormality
* Subject practicing windsurfing (whatever the level of practice (leisure or competition))

Exclusion Criteria:

* Subjects < 18 years old
* Pregnant woman
* Inability to consent
* Taking any of the following: oral or inhaled Beta 2 short-acting or long-acting mimetics, oral or inhaled corticosteroids, oral anti-leukotrienes.
* Abnormalities in the resting ECG pattern

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC in L) at rest. | 1 day
  spirometry at rest

SECONDARY OUTCOMES:
Forced Expiratory Volume | 1 day
  FEV1 (in L)
Peak Flow | 1 day
  PF (peak flow in L/s)
mean flow rates | 1 day
  mean expiratory flow rates in L/ s at 75%, 50% and 25% of FVC (MEF 75, MEF 50, MEF 25).
maximal ventilation | 1 day
  VE (ventilation in L/min)
carbon dioxide production | 1 day
  VCO2 ( in L/min)
oxygen consumption | 1 day
  VO2 ( in L/min)
tidal volume | 1 day
  VT (in L)
breathing frequency | 1 day
  RF (in breaths/min)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Agnes Giroux-Metges, Pr, Principal Investigator — CHRU de Brest
Locations (1):
- University hospital, Brest, France